CLINICAL TRIAL: NCT01688986
Title: Environmental Polymorphisms Registry Health and Exposures Survey
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120194; 12-E-0194
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2016-11-22

CONDITIONS: Diabetes; Heart Disease; Asthma
Keywords: Complex Disease; DNA Biorepository; Genotype-Phenotype Correlation; Genetics; Environmental Factors
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The Environmental Polymorphisms Registry (EPR) Health and Exposure Survey is designed to gather health, family history of disease, environmental exposures and lifestyle data on adult EPR subjects. The EPR is a registry established to collect and store DNA samples from 20,000 volunteers from North Carolina and to serve as a resource to scientist investigating genotype-driven translational research of chronic conditions. Under this new protocol, we will administer a health and exposures survey to all EPR subjects. The information collected in the survey will be used to better characterize the EPR population thus making it more useful to NIEHS researchers. The survey contains approximately 200 questions. Data from the survey will help researchers develop hypotheses, design follow-up studies, and select appropriate subjects.

The survey will be administered to EPR subjects using a modified version of the Dillman Total Design Method (TDM) for surveys. This method requires following specific time-dependent steps for survey administration that incorporate both self- and phone administration and other types of phone and mail contact. The goal of TDM is to maximize subject response rates.

DETAILED DESCRIPTION:
The Environmental Polymorphisms Registry (EPR) Health and Exposure Survey is designed to collect health, family history of disease, environmental exposures and lifestyle data on EPR participants. The EPR was established to collect and store DNA specimens from 20,000 participants and to serve as a resource for scientists investigating genotype-driven translational research of chronic health conditions. Under this protocol, we will administer the approximately 200 question Health and Exposure Survey to EPR participants. The information will be used to better characterize the EPR population, thus making it more useful in answering research questions related to gene-environment interactions. Data from the survey will help researchers to advance clinical research by developing new ways of preventing, diagnosing, and treating common diseases such as cardiovascular disease, asthma, and diabetes.

During Phases I and II, the survey was administered to EPR participants using a modified version of the Dillman Total Design Method (TDM) for surveys. This method requires following specific steps for survey administration that incorporate web-based, paper and phone administration. The rationale for using the TDM is to maximize participant response rates. During Phase III, the survey may be distributed to new EPR participants (e.g., those who were not enrolled in the EPR at the time of the Phase I and II survey administrations) for self-administration at the time of enrollment.

Investigators may select and contact participants for follow-up studies based upon health, exposure, or disease status information; this includes responses to the EPR Health and Exposure Survey. Participation in follow-up studies is completely voluntary. Participants can decide at the time they are contacted if they would like to enroll in the follow-up study. Their decision whether or not to participate in a follow-up study will not affect their participation in the EPR.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

There are no clinical exclusion criteria for this Survey. All subjects will be administered the Survey regardless of having clinical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9000 (Actual)
Dates: Start 2012-08-25; Study Completion 2016-11-22

CONTACTS AND LOCATIONS:
Overall Officials: Shepherd H Schurman, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- [Derived] Whitehead GS, Hussain S, Fannin R, Trempus CS, Innes CL, Schurman SH, Cook DN, Garantziotis S. TLR5 Activation Exacerbates Airway Inflammation in Asthma. Lung. 2020 Apr;198(2):289-298. doi: 10.1007/s00408-020-00337-2. Epub 2020 Feb 14. PMID 32060608